CLINICAL TRIAL: NCT05497167
Title: Development and Evaluation of "Period Kits" for Adolescents With Intellectual and Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00002861
Record Dates: First submitted 2022-07-22; First posted 2022-08-11 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Autistic Spectrum Disorder; Patient Empowerment; Menstrual Discomfort
Keywords: menarche; autism; intellectual and developmental disability; patient education; period resources
MeSH Terms: conditions — Autism Spectrum Disorder; Patient Participation; Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Subjects will be patients with intellectual and developmental disability who have not yet had menarche.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Period Kit (Experimental): This is a single arm interventional study wherein the subjects enrolled will all participate in the study in the same way by being asked to answer pre-study survey questions concerning their attitudes towards menarche, receiving a period kit to explore on their own for two weeks, and then being asked to answer post-study survey questions.
  Interventions: Other: Period Kit

INTERVENTIONS:
Other: Period Kit — This is a single arm interventional study wherein the subjects enrolled will all participate in the study in the same way by being asked to answer pre-study survey questions concerning their attitudes towards menarche, receiving a period kit to explore on their own for two weeks, and then being asked to answer post-study survey questions.

SUMMARY:
This study will involve the development, distribution, and evaluation of "period kits" for pre-menarchal adolescents with intellectual and cognitive disabilities (IDD) (e.g., autism spectrum disorder and Down syndrome) in relieving stress and augmenting sense of preparedness regarding imminent pubertal changes.

DETAILED DESCRIPTION:
Overview of procedures:

1. Screening phone call with parent/guardian (10-15 minutes)
2. Initial study visit and pre-study survey, on Zoom with parent/guardian and minor (60 minutes)
3. In-person period kit distribution at the Center for Children with Special Needs with parent/guardian and minor (5-10 minutes)
4. Two-week interlude for participants to experiment with kit components
5. Final study visit and post-study survey, on Zoom with parent/guardian and minor (60 minutes)

This study will involve distributing and evaluating the efficacy of "period kits" for approximately 15-25 pre-menarchal participants and parent/guardian pairs. Study participants will be selected by convenience sampling for adolescents under 18 years of age with imminent medical appointments at the Center for Children with Special Needs (CCSN) at Tufts; if more participants are needed, Dr. Crehan will assist in recruitment from other networks (e.g., through social media posts on Facebook and Instagram, and posting on the Crehan lab website at https://sites.tufts.edu/crehanlab/).

If contacted participants express interest to participate, the study team will engage with them in a screening phone call to further discuss the study, as well as verify eligibility and CCSN appointment date and time so that the initial Zoom study visit may be scheduled on a date preceding the CCSN appointment. After this phone call, participants will be sent a Visit 1 invitation email with Zoom information for this first study visit.

At the initial study visit, members of the study team will meet prospective on Zoom at the time scheduled in the screening phone call. Team members will explain the study design, reinforce that participation is optional, and obtain consent/assent from each adolescent participant and respective parent/guardian. Study team members will briefly interview the participating minor and parent/guardian and receive verbal responses. Then, study team members will administer a brief Qualtrics pre-study survey (15 minutes) for completion by each participant's parent/guardian on their own device. Finally, during the same visit, study team members will go over all contents of the period kit, ensuring to answer any questions that may arise. The study team will then confirm the time of the participant's upcoming CCSN appointment, reiterate that the participant will be given a period kit at the CCSN immediately following the appointment, and arrange a visit after a two-week trial period to discuss kit efficacy in mitigating any puberty- and menstruation-related concerns and anxieties.

Period kit components will constitute the following:

1. Period management resources for practice with sensory stimuli, including:

   a. Appropriately sized pads, tampons, and period underwear
2. Menstruation-related social story b. Includes easily interpretable graphics on how to appropriately and hygienically manage menstruation, as well as terminology with which to refer to relevant anatomy and respective functions
3. Illustrated resource list, including:

   c. Evidence-based free period tracking apps d. Evidence-based puberty-related books e. Hormonal menstrual suppression: indication as a period management option, and suggestion to discuss, if interested, with a pediatrician f. Symptom management suggestions: e.g., over-the-counter pain medications, exercise, and heating pads
4. Zippered pouch encasing all aforementioned supplies, for convenient handling and use by study participants. Participants will be able to keep all supplies after participation.

After the two-week trial period, the study team will meet with all participants again on Zoom to ask questions to the participating minor and parent/guardian and receive verbal responses. The study team will then administer the post-study survey (15 minutes) on Qualtrics to evaluate how kit components may have impacted families' anxiety levels and sense of knowledge and preparedness concerning menstruation and other imminent developmental changes. The survey will be conducted online, with results only accessible by study team members.

A thematic analysis will be performed for qualitative evaluation of all collected data; questionnaires will be margin coded to identify unique and recurrent themes using a modified grounded theory approach in an iterative process. Content analysis will be used to identify themes across study participants. Discrepancies in coding will be resolved using a constant comparison and consensus approach. All responses will be imported into a web-based software program (NVivo) to facilitate the organization and analyses of this qualitative data.

ELIGIBILITY:
Inclusion Criteria:

1. Minors from 5 to 17 years of age
2. Those with the capacity to eventually menstruate but who have not yet had a menstrual period
3. Those with an Intellectual and Developmental Disability (IDD), defined here using DSM diagnostic labels: autism spectrum disorder, Global Developmental Delay, Unspecified Neurodevelopmental Disorder (which includes Down Syndrome and fragile-X)

Exclusion Criteria:

1. Those that do not meet any of the aforementioned criteria
2. Minors who are:

   i) married, widowed, divorced; or ii) the parent of a child; or iii) a member of any of the armed forces; or iv) pregnant or believes herself to be pregnant; or v) living separate and apart from his/her parent or legal guardian, and is managing his/her own financial affairs
3. Wards of the state and/or children at risk of becoming wards of the state
4. Non-English speakers

Ages: 5 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Number of participants who report feeling more comfortable and/or prepared for menstruation after period kit exploration | 12 months
  The aim of the study is to develop, optimize, and evaluate the efficacy of a "period kit" for adolescents with cognitive disability and their families. The purpose of the kit is to familiarize and educate this population about menstruation and other puberty-related changes, ideally prior to the first menstrual period. Response to this kits will inform future work on whether these materials are helpful for medical care teams to provide education and resources for patients with intellectual and developmental disabilities. The study outcome will be measured by the number of subjects who report feeling more comfortable and/or prepared for menstruation after period kit exploration, based on questionnaire responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogan V, Lake JK, Tint A, Weiss JA, Lunsky Y. Tracking health care service use and the experiences of adults with autism spectrum disorder without intellectual disability: A longitudinal study of service rates, barriers and satisfaction. Disabil Health J. 2017 Apr;10(2):264-270. doi: 10.1016/j.dhjo.2016.11.002. Epub 2016 Nov 22. PMID 27899267
- [Background] Chiri G, Warfield ME. Unmet need and problems accessing core health care services for children with autism spectrum disorder. Matern Child Health J. 2012 Jul;16(5):1081-91. doi: 10.1007/s10995-011-0833-6. PMID 21667201
- [Background] Muskat B, Burnham Riosa P, Nicholas DB, Roberts W, Stoddart KP, Zwaigenbaum L. Autism comes to the hospital: the experiences of patients with autism spectrum disorder, their parents and health-care providers at two Canadian paediatric hospitals. Autism. 2015 May;19(4):482-90. doi: 10.1177/1362361314531341. Epub 2014 May 8. PMID 24811967